CLINICAL TRIAL: NCT00615472
Title: Intravenous General Anesthesia Versus Inhalational General Anesthesia in Parkinson's Disease
Brief Title: Intravenous Versus Inhalational Anesthesia in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Eric J. Heyer, MD, PhD, Professor of Clinical Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AAAA4885
Record Dates: First submitted 2008-01-09; First posted 2008-02-14 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Deep brain stimulation (DBS); Subthalamic Nucleus; Total Intravenous Anesthesia; Inhalational Anesthesia
MeSH Terms: conditions — Parkinson Disease | interventions — Isoflurane; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Inhaled Anesthesia - isoflurane
  Interventions: Drug: Isoflurane
- Group 2 (Experimental): Intravenous Anesthesia - propofol, remifentanil
  Interventions: Drug: Remifentanil; Drug: Propofol

INTERVENTIONS:
Drug: Isoflurane — Group 1 Inhaled anesthesia Patients will be maintained on 50% oxygen in air and isoflurane 0 to 4%, titrated as needed to maintain a standard blood pressure (standard practice). If needed, muscle relaxation will be provided by additional boluses or an infusion of mivacurium (4-10 ug/kg/min).
  Other Names: Forane
  Arms: Group 1
Drug: Remifentanil — Group 2 Intravenous anesthesia Patients will be ventilated with 50% oxygen in air. Patients will receive continuous propofol infusion 0.05 mg/kg-min to 0.15 mg/kg-min titrated as needed; and remifentanil (ultra-short acting narcotic) 0.1 ug/kg-min to 0.5 ug/kg-min. These will be titrated as needed to maintain a standard blood pressure. Both infusions will be turned off at the end of the procedure. If needed, muscle relaxation will be provided by additional boluses or an infusion of mivacurium (4-10 ug/kg/min).
  Other Names: Ultiva
  Arms: Group 2
Drug: Propofol — Group 2 Intravenous anesthesia Patients will be ventilated with 50% oxygen in air. Patients will receive continuous propofol infusion 0.05 mg/kg-min to 0.15 mg/kg-min titrated as needed; and remifentanil (ultra-short acting narcotic) 0.1 ug/kg-min to 0.5 ug/kg-min. These will be titrated as needed to maintain a standard blood pressure. Both infusions will be turned off at the end of the procedure. If needed, muscle relaxation will be provided by additional boluses or an infusion of mivacurium (4-10 ug/kg/min).
  Other Names: Diprivan
  Arms: Group 2

SUMMARY:
Parkinson's disease is a common progressive degenerative disease affecting 3% of all patients over the age of 65. Given their age and frailty, these patients frequently require surgical procedures with general anesthesia. However, after surgery, patients with Parkinson's disease have longer hospital stays and a greater chance of not returning to independent living compared to age-matched controls (Berman MF, unpublished data). In part, this is due to a higher rate of post-operative delirium, which had an incidence of 60% in this population in one study. There is anecdotal evidence from neurologists specializing in movement disorder suggesting that there is also significant deterioration in parkinsonian motor symptoms and cognition lasting for months or years following surgery and anesthesia. The basis for this deterioration is unknown. We hypothesize that these problems are caused by particular medications used during inhaled anesthesia for surgical procedures.

DETAILED DESCRIPTION:
We will compare the groups in terms of postoperative delirium, and cognitive and motor function changes. Patients randomized to an inhaled anesthetic will receive a standard anesthetic mix: an inhaled anesthetic with intravenous agents for rapid induction of anesthesia, narcotics for postoperative pain relief, and muscle relaxation. Patients randomized to IV anesthesia will receive a continuous infusion of propofol and remifentanil (ultrashort acting narcotic) instead of the inhalation anesthetics during the maintenance phase of the anesthetic. Other components of the anesthetic will be the same as in the "inhaled anesthetic" group.

We hypothesize that:

1. Patients with Parkinson's disease will have less postoperative delirium and less prolonged cognitive and motor changes after total intravenous anesthesia than following inhaled anesthesia.
2. Apolipoprotein E4 (Apo E4) allele will be associated with postoperative cognitive dysfunction in Parkinsonian patients

To test our hypotheses we will:

1. Randomize patients with Parkinson's disease having surgery for implantation of current generator for subthalamic stimulator to receive either a total intravenous anesthetic or an inhaled anesthetic.
2. Compare these two groups of patients for incidence of postoperative delirium and the degree of postoperative cognitive and motor dysfunction.
3. Test for an association between the (Apo E4) allele and postoperative cognitive change. A buccal sampling or cheek cell sampling method will be employed to obtain DNA for genotyping of the Apo E allele.

During the procedure, maintenance of anesthesia will differ for the two groups:

Group 1 Inhaled anesthesia: Patients will be maintained on oxygen and isoflurane 0 to 4%, titrated as needed to maintain a standard blood pressure (standard practice).

Group 2 Intravenous anesthesia: Patients will be ventilated with 50% oxygen in air. Patients will receive continuous propofol infusion 0.05 mg/kgmin to 0.15 mg/kgmin titrated as needed; and remifentanil (ultrashort acting narcotic) 0.1 ug/kgmin to 0.5 ug/kgmin. These will be titrated as needed to maintain a standard blood pressure. Both infusions will be turned off at the end of the procedure.

Testing of Motor and Cognitive Status. Patients who participate in the study will be given a mental status examination, tests of Parkinsonian motor symptoms, and tests of cognitive function in the preoperative period before implantation of the subthalamic electrodes and implantation of current generators. Subsets of these tests will be performed several times postoperatively (1 month and 4 months)

Implantation of Electrode (Stage I sedation anesthesia) Full testing will be done in the preoperative period. Patients are generally kept in the hospital overnight and discharged the following day. Mental status will be rechecked by the MMSE in the recovery room postoperatively .

Patients will be contacted by telephone to have their mental status assessed by telephone using using two well known examinations (Telephone Interview for Cognitive Status (TICS) and Centers for Disease Control and Prevention Health-Related Quality-of-Life 14Item Measure (CDC HRQOL14)) and a series of questions investigating how well patients are able to perform activities of daily living (ADLs) and instrumental activities of daily living (IADLs). These tests will be given at two time points, once before the surgery and then one month after surgery. We will look for changes in quality of life that may correlate with neuropsychometric test performance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease with bilateral deep brain stimulation surgery indicated as treatment

Exclusion Criteria:

* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-10; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Heyer, M.D., Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia Unviversity, Deparment of Anesthesiology, New York, New York, United States

REFERENCES:
- [Background] Corder EH, Saunders AM, Strittmatter WJ, Schmechel DE, Gaskell PC, Small GW, Roses AD, Haines JL, Pericak-Vance MA. Gene dose of apolipoprotein E type 4 allele and the risk of Alzheimer's disease in late onset families. Science. 1993 Aug 13;261(5123):921-3. doi: 10.1126/science.8346443.
- [Background] Friedman G, Froom P, Sazbon L, Grinblatt I, Shochina M, Tsenter J, Babaey S, Yehuda B, Groswasser Z. Apolipoprotein E-epsilon4 genotype predicts a poor outcome in survivors of traumatic brain injury. Neurology. 1999 Jan 15;52(2):244-8. doi: 10.1212/wnl.52.2.244. PMID 9932938
- [Background] Brandt R, Spencer M, Folstein M: The Telephone Interview for Cognitive Status. Neuropsychiatry, Neuropsychology, and Behavioral Neurology 1:111-117, 1988.
- [Background] Culley DJ, Yukhananov RY, Baxter MB, Crosby G: Longerterm cognitive performance after general anesthesia in aged rats. J Neurosurg Anesthesiol 12:395 (abstract 325), 2000.
- [Background] Golden WE, Lavender RC, Metzer WS. Acute postoperative confusion and hallucinations in Parkinson disease. Ann Intern Med. 1989 Aug 1;111(3):218-22. doi: 10.7326/0003-4819-111-3-218. PMID 2751180
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Newman MF, Croughwell ND, Blumenthal JA, Lowry E, White WD, Spillane W, Davis RD Jr, Glower DD, Smith LR, Mahanna EP, et al. Predictors of cognitive decline after cardiac operation. Ann Thorac Surg. 1995 May;59(5):1326-30. doi: 10.1016/0003-4975(95)00076-w. PMID 7733762
- [Background] Patten D, Foxon GR, Martin KF, Halliwell RF. An electrophysiological study of the effects of propofol on native neuronal ligand-gated ion channels. Clin Exp Pharmacol Physiol. 2001 May-Jun;28(5-6):451-8. doi: 10.1046/j.1440-1681.2001.03469.x. PMID 11380521
- [Background] Pepper PV, Goldstein MK. Postoperative complications in Parkinson's disease. J Am Geriatr Soc. 1999 Aug;47(8):967-72. doi: 10.1111/j.1532-5415.1999.tb01292.x. PMID 10443858
- [Background] Ruberg M, Ploska A, Javoy-Agid F, Agid Y. Muscarinic binding and choline acetyltransferase activity in Parkinsonian subjects with reference to dementia. Brain Res. 1982 Jan 28;232(1):129-39. doi: 10.1016/0006-8993(82)90615-1. PMID 7055689
- [Background] Spreen O, Strauss E: A compendium of Neuropsychological tests. New York, Oxford University Press, 1998, ed second.
- [Background] van Laar T, Jansen EN, Essink AW, Neef C, Oosterloo S, Roos RA. A double-blind study of the efficacy of apomorphine and its assessment in 'off'-periods in Parkinson's disease. Clin Neurol Neurosurg. 1993 Sep;95(3):231-5. doi: 10.1016/0303-8467(93)90128-4. PMID 8242966
- [Background] Violet JM, Downie DL, Nakisa RC, Lieb WR, Franks NP. Differential sensitivities of mammalian neuronal and muscle nicotinic acetylcholine receptors to general anesthetics. Anesthesiology. 1997 Apr;86(4):866-74. doi: 10.1097/00000542-199704000-00017. PMID 9105231
- [Background] Williams-Russo P, Sharrock NE, Mattis S, Szatrowski TP, Charlson ME. Cognitive effects after epidural vs general anesthesia in older adults. A randomized trial. JAMA. 1995 Jul 5;274(1):44-50. PMID 7791257
- [Background] Ali HH, Savarese JJ, Embree PB, Basta SJ, Stout RG, Bottros LH, Weakly JN. Clinical pharmacology of mivacurium chloride (BW B1090U) infusion: comparison with vecuronium and atracurium. Br J Anaesth. 1988 Nov;61(5):541-6. doi: 10.1093/bja/61.5.541. PMID 2905143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled only a few patients. Our neurocognitive battery was too hard for patients to get through. Therefore, the study was stopped.
Groups:
- Inhaled Anesthesia: Inhaled Anesthesia - isoflurane
- Intravenous Anesthesia: Intravenous Anesthesia - propofol, remifentanil
Period: Overall Study
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia
Started | 30 | 28
Completed | 30 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients had neuropsychometric analysis before and after procedure.
Groups:
- Inhaled Anesthesia: Inhaled Anesthesia - isoflurane
  Isoflurane: Group 1 Inhaled anesthesia Patients will be maintained on 50% oxygen in air and isoflurane 0 to 4%, titrated as needed to maintain a standard blood pressure (standard practice). If needed, muscle relaxation will be provided by additional boluses or an infusion of mivacurium (4-10 ug/kg/min).
- Intravenous Anesthesia: Intravenous Anesthesia - propofol, remifentanil
  Remifentanil: Group 2 Intravenous anesthesia Patients will be ventilated with 50% oxygen in air. Patients will receive continuous propofol infusion 0.05 mg/kg-min to 0.15 mg/kg-min titrated as needed; and remifentanil (ultra-short acting narcotic) 0.1 ug/kg-min to 0.5 ug/kg-min.
  Propofol: Group 2 Intravenous anesthesia Patients will be ventilated with 50% oxygen in air. Patients will receive continuous propofol infusion 0.05 mg/kg-min to 0.15 mg/kg-min titrated as needed
- Total: Total of all reporting groups
Arm/Group | Inhaled Anesthesia | Intravenous Anesthesia | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 28 | 58
Age, Continuous [Mean (Full Range); unit: years] | 67 [65 to 72] | 69 [66 to 73] | 68 [65 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved Postoperative Delirium and Cognitive and Motor Changes
Description: A battery/Questionnaire of neuropsych examinations is given to the subjects to measure improvement based on change of scores and standard deviation. The battery consists of questions regarding delirium, cognitive and motor changes and yields a combination assessment of all 3 elements.
Time Frame: Four months
Measure: Number; unit: participants
Groups:
- Group 2: Intravenous Anesthesia - propofol, remifentanil
  Remifentanil: Group 2 Intravenous anesthesia Patients will be ventilated with 50% oxygen in air. Patients will receive continuous propofol infusion 0.05 mg/kg-min to 0.15 mg/kg-min titrated as needed; and remifentanil (ultra-short acting narcotic) 0.1 ug/kg-min to 0.5 ug/kg-min.
  Propofol: Group 2 Intravenous anesthesia Patients will be ventilated with 50% oxygen in air. Patients will receive continuous propofol infusion 0.05 mg/kg-min to 0.15 mg/kg-min titrated as needed; and remifentanil (ultra-short acting narcotic) 0.1 ug/kg-min to 0.5 ug/kg-min.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 30 | 28
participants | 6 | 5

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No